CLINICAL TRIAL: NCT06807346
Title: A Randomized, Triple-blind, Placebo-controlled Trial Evaluating the Efficacy of the Study Product on Overall Cognitive Function in Children
Brief Title: Evaluating the Efficacy of the Study Product on Overall Cognitive Function in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SmartyPants Vitamins Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24SVCFS01
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-01

CONDITIONS: Cognition
Keywords: Cognition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kids Plus Multi & Omegas (Experimental): Kids Plus Multi & Omega is a dietary supplement contains a mixture of vitamins, minerals, and omega-3 fatty acids.
  Interventions: Dietary Supplement: Kids Plus Multi & Omega
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Kids Plus Multi & Omega — Participants will be instructed to take two gummies of Kids Plus Multi and Omegas with or without food once daily for the duration of the study starting on Day 1 with a recommendation to consume in the morning for consistency.
  Arms: Kids Plus Multi & Omegas
Dietary Supplement: Placebo — Participants will be instructed to take two gummies of placebo with or without food once daily for the duration of the study starting on Day 1 with a recommendation to consume in the morning for consistency.
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of Kids Plus Multi & Omega dietary supplement on cognitive function in children after 49 days of supplementation. The main question it aims to answer is:

Is there a difference in change in individual cognitive domains between Kids Plus Multi & Omega and placebo?

Participants will be asked to consume Kids Plus Multi & Omega or placebo and complete various cognitive assessment tests throughout the duration of the study.

DETAILED DESCRIPTION:
The investigational product, Kids Plus Multi & Omega dietary supplement contains a mixture of vitamins, minerals, and omega-3 fatty acids. Emerging evidence reports the positive effects of micronutrient supplementation on cognitive performance among school-aged children. However, there is still limited evidence on the efficacy of multiple micronutrient supplementation on other aspects of cognitive function in children. Therefore, the objective of this randomized, triple-blind placebo-controlled clinical trial is to evaluate the efficacy of Kids Plus Multi & Omega dietary supplement on cognitive function in children after 49 days of supplementation. Overall cognitive function as well as cognitive domains related to focus, memory, learning and cognitive flexibility will be assessed using the National Institutes of Health (NIH) Toolbox Cognition Battery.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females 4-17 years of age, inclusive
2. Females of child-bearing potential must have a negative screening urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:

   * Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
   * Double-barrier method
   * Intrauterine devices
   * Non-heterosexual lifestyle and agrees to use contraception if planning on changing to heterosexual partner(s)
   * Vasectomy of partner at least 6 months prior to screening
   * Abstinence and agrees to use contraception if planning to become sexually active during the study
3. Enrolled in and currently attending school at baseline and for the duration of the study period
4. Willing to complete evaluations, measurements, questionnaires and diaries during each clinic visit
5. Agrees to avoid eating or moderate-vigorous exercise for one hour prior to clinic visits
6. Agrees to maintain current lifestyle habits (diet, physical activity, medications, supplements, and sleep) as much as possible throughout the study and avoid taking new supplements
7. A care provider who can reliably bring the participant to all study visits; the participant's primary caregiver must be willing and able to complete the questionnaires as needed for all visits
8. The child and the child's parent(s) or legal guardian(s) have given voluntary, written, informed assent and consent, respectively, for their child to participate in the study
9. Healthy as determined by medical history as assessed by Qualified Investigator (QI)

Exclusion Criteria:

1. Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
2. Allergy, sensitivity, or intolerance to the investigational product or placebo ingredients
3. Previous diagnosis or treatment of a significant neuropsychological condition and/or cognitive impairment (e.g., Schizophrenia, bipolar disorder, post-traumatic stress disorder, brain injury, neurodegenerative disease, infections, insomnia, depression, epileptic or other seizure-related disorders) that could interfere with study participation as assessed by the QI
4. Unable to communicate or cooperate due to language problems, learning disability, poor mental development, or impaired cerebral functions as assessed by the QI
5. Previous diagnosis of Attention-deficit hyperactivity disorder (ADHD)
6. Previous diagnosis of visual (including color blindness/weakness) or hearing impairment that may impact task performance as assessed by the QI
7. Currently experiencing major social/family stressors as confirmed by the child's parent or legal guardian (s)
8. History or presence of a clinically relevant cardiac, renal, hepatic, endocrine (including diabetes mellitus), pulmonary, biliary, gastrointestinal condition which affects absorption, or pancreatic disorders, as assessed by the QI
9. Cancer, except skin basal cell carcinoma completely excised with no chemotherapy or radiation with a follow up that is negative. Volunteers with cancer in full remission for more than five years after diagnosis are acceptable
10. Individuals with an autoimmune disease or are immune compromised
11. Use of cannabinoid, tobacco or nicotine-containing products, or alcohol consumption
12. Alcohol or drug abuse within the last 12 months
13. Current use of prescribed and/or over-the-counter (OTC) medications, supplements, and/or consumption of food/drinks that may impact the efficacy of the investigational product (Sections 7.3.1 and 7.3.2)
14. Employees/children of employees of study sponsor or research organization
15. Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
16. Parent or guardian who are unable to give informed consent
17. Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 4 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2025-05-06 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
The difference in change in individual cognitive domains between Kids Plus Multi and Omega and placebo | Day 0 (baseline) to 28
  The difference in change in individual cognitive domains as assessed by the NIH Toolbox Cognition tests from baseline at Day 28 between Kids Plus Multi and Omega and placebo
The difference in change in individual cognitive domains between Kids Plus Multi and Omega and placebo | Day 0 (baseline) to 49
  The difference in change in individual cognitive domains as assessed by the NIH Toolbox Cognition tests from baseline at Day 49 between Kids Plus Multi and Omega and placebo

SECONDARY OUTCOMES:
The difference in change in Total Cognition Composite score (for children aged 7+ years) or Early Childhood Composite score (for children aged 4-6 years) between Kids Plus Multi and Omega and placebo | Day 0 (baseline) to 28
  The difference in change in Total Cognition Composite score (for children aged 7+ years) or Early Childhood Composite score (for children aged 4-6 years) as assessed by the NIH Toolbox Cognition tests from baseline at Day 28 between Kids Plus Multi and Omega and placebo
The difference in change in Total Cognition Composite score (for children aged 7+ years) or Early Childhood Composite score (for children aged 4-6 years) between Kids Plus Multi and Omega and placebo | Day 0 (baseline) to 49
  The difference in change in Total Cognition Composite score (for children aged 7+ years) or Early Childhood Composite score (for children aged 4-6 years) as assessed by the NIH Toolbox Cognition tests from baseline at Day 49 between Kids Plus Multi and Omega and placebo
The difference in change in quality of life between Kids Plus Multi and Omega and placebo | Day 0 (baseline) to 28
  The difference in change in quality of life as assessed by the KINDL-R questionnaire between Kids Plus Multi and Omega and placebo from baseline at Day 28.
The difference in change in quality of life between Kids Plus Multi and Omega and placebo | Day 0 (baseline) to 49
  The difference in change in quality of life as assessed by the KINDL-R questionnaire between Kids Plus Multi and Omega and placebo from baseline at Day 49
The difference in change in stress between Kids Plus Multi and Omega and placebo | Day 0 (baseline) to 28
  The difference in change in stress as assessed by Perceived Stress Scale for Children (PSS-C) between Kids Plus Multi and Omega and placebo from baseline at Day 28. The PSS-C has a scale range from 0-39 with higher scores indicating higher stress levels.
The difference in change in stress between Kids Plus Multi and Omega and placebo | Day 0 (baseline) to 49
  The difference in change in stress as assessed by Perceived Stress Scale for Children (PSS-C) between Kids Plus Multi and Omega and placebo from baseline at Day 49. The PSS-C has a scale range from 0-39 with higher scores indicating higher stress levels.

OTHER OUTCOMES:
Incidence of post-emergent adverse events (AE) | Day 0 (baseline) to 49
  Incidence of post-emergent adverse events (AE) between Kids Plus Multi and Omega and placebo
Clinically relevant changes in blood pressure (BP) after supplementation | Day 0 (baseline) to 49
  Clinically relevant changes in blood pressure (BP) after supplementation with Kids Plus Multi and Omega
Clinically relevant changes in heart rate (HR) after supplementation | Day 0 (baseline) to 49
  Clinically relevant changes in heart rate (HR) after supplementation with Kids Plus Multi and Omega.

CONTACTS AND LOCATIONS:
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No